CLINICAL TRIAL: NCT01807026
Title: A Safety, Pharmacokinetic, and Pharmacodynamic Study of LY2886721 in Healthy Subjects and Patients Diagnosed With Alzheimer's Disease
Brief Title: A Study of LY2886721 in Healthy Participants and Participants Diagnosed With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 15107; I4O-EW-BACX (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer Disease; Healthy Volunteers
MeSH Terms: conditions — Alzheimer Disease | interventions — N-(3-(2-amino-4a,5,7,7a-tetrahydro-4H-furo(3,4-d)(1,3)thiazin-7a-yl)-4-fluorophenyl)-5-fluoropicolinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort A: 70 mg LY2886721 (Experimental): Participants with Alzheimer's disease received a single, 70-milligrams (mg) (1 capsule), oral dose of LY2886721.
  Interventions: Drug: LY2886721
- Cohort A: Placebo (Placebo Comparator): Participants with Alzheimer's disease received a single, oral dose of LY2886721-matching placebo (1 capsule).
  Interventions: Drug: Placebo
- Cohort B: 70 mg LY2886721 (Experimental): Healthy participants received a single, 70-mg (1 capsule), oral dose of LY2886721.
  Interventions: Drug: LY2886721
- Cohort B: Placebo (Placebo Comparator): Healthy participants received a single, oral dose of LY2886721-matching placebo (1 capsule).
  Interventions: Drug: Placebo
- Cohort C: 280 mg LY2886721 (Experimental): Healthy participants received a single, 280-mg (4 x 70 mg capsules), oral dose of LY2886721.
  Interventions: Drug: LY2886721
- Cohort C: Placebo (Placebo Comparator): Healthy participants received a single, oral dose of LY2886721-matching placebo (4 capsules).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2886721
  Arms: Cohort A: 70 mg LY2886721; Cohort B: 70 mg LY2886721; Cohort C: 280 mg LY2886721
Drug: Placebo
  Arms: Cohort A: Placebo; Cohort B: Placebo; Cohort C: Placebo

SUMMARY:
This study is being done for the following reasons:

To determine the safety of LY2886721 and any side effects that may be associated with it and to see how much of the study drug is in the blood and the cerebrospinal fluid (CSF) when one dose is given to healthy participants and participants diagnosed with Alzheimer's disease. It will also look at how safe and tolerable the study drug is when given to healthy participants in higher doses.

This research study is being conducted in three groups, referred to as Groups (Cohorts) A, B, or C.

Group A will enroll participants with Alzheimer's disease while Groups B and C will enroll healthy participants.

For Group A or B, participation in this research study could last up to 34 days. For Group C, participation could last up to 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants have a body mass index (BMI) of 19 to 32 kilograms per square meter (kg/m^2), inclusive, at screening. There are no restrictions on BMI in participants diagnosed with Alzheimer's disease.
* Healthy participants should not be taking any concomitant medications. For participants with Alzheimer's disease, concomitant medications will be determined by the investigator in consultation with the Lilly clinical pharmacologist on an individual basis.

Cohort A:

* Participants are defined as otherwise healthy males or females as determined by medical history and physical examination, and a diagnosis of Alzheimer's disease and must be at least 45 years of age.
* Meets National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable Alzheimer's disease, as determined by a clinician approved by the sponsor or designee.
* Mini Mental State Examination (MMSE) score of 16 through 28 at screening.
* Modified Hachinski Ischemia Scale (MHIS) score of <4.
* Capable of understanding and signing their own informed consent, in the opinion of the investigator, or if the participant has a Legally Authorized Representative (LAR), then the LAR must be capable of understanding and signing the assent form, and the participant may or may not sign the informed consent, as to be determined by the investigator.
* If receiving concurrent treatment with an acetylcholinesterase inhibitor (AChEI) and/or memantine, the participant has been on a stable dose for at least 4 weeks before Day 1. Dosing must remain stable throughout the study. Note: If a participant has recently stopped ACHEIs and/or memantine, he or she must have discontinued treatment for at least 4 weeks before Day 1.

Exclusion Criteria:

* Have an abnormality in the 12-lead electrocardiogram (ECG).
* Have abnormal blood pressure.
* Have abnormal thyroid function as reflected by thyroid stimulating hormone (TSH) values outside of the normal range.
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Have had multiple episodes of head trauma, or have a history within the last 5 years of a serious infectious disease affecting the brain.
* Have chronic hepatic disease.
* Have evidence or history of significant active bleeding or a coagulation disorder.
* Cohort A: have any neurological disorders other than Alzheimer's disease.
* For healthy participants (Cohorts B and C) only: Use or intend to use over the- counter or prescription medication, including herbal medications within 14 days prior to dosing or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort A: Placebo | Cohort B: 70 mg LY2886721 | Cohort B: Placebo | Cohort C: 280 mg LY2886721 | Cohort C: Placebo
Started | 10 | 2 | 10 | 2 | 9 | 3
Received at Least One Dose of Study Drug | 10 | 2 | 10 | 2 | 9 | 3
Completed | 10 | 2 | 10 | 2 | 9 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Cohort A: 70 mg LY2886721: Participants with Alzheimer's disease received a single, 70-mg (1 capsule), oral dose of LY2886721.
- Total: Total of all reporting groups
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort A: Placebo | Cohort B: 70 mg LY2886721 | Cohort B: Placebo | Cohort C: 280 mg LY2886721 | Cohort C: Placebo | Total
Number analyzed (Participants) | 10 | 2 | 10 | 2 | 9 | 3 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (12.6) | 67.0 (18.4) | 59.3 (6.8) | 54.5 (3.5) | 29.3 (11.3) | 21.3 (0.6) | 51.8 (20.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 5 | 1 | 1 | 0 | 14
  Male | 4 | 1 | 5 | 1 | 8 | 3 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 10 | 2 | 10 | 2 | 8 | 3 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 2 | 10 | 2 | 9 | 3 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Area Under the Curve Extrapolated to Infinity (AUC0-∞) of Plasma LY2886721
Description: AUC0-∞ following administration of a single dose of 70 or 280 mg LY2886721.
Time Frame: Predose through 96 hours after administration of study drug
Population: Participants who received at least one dose of LY2886721 and with evaluable plasma LY2886721-concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*h/mL)
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort B: 70 mg LY2886721 | Cohort C: 280 mg LY2886721
Number analyzed (Participants) | 10 | 10 | 9
nanograms*hours/milliliter (ng*h/mL) | 2800 (25) | 2580 (20) | 10500 (22)

2. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Plasma LY2886721
Description: Cmax following administration of a single dose of 70 or 280 mg LY2886721.
Time Frame: Predose through 96 hours after administration of study drug
Population: Participants who received at least one dose of LY2886721 and with evaluable plasma LY2886721-concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort B: 70 mg LY2886721 | Cohort C: 280 mg LY2886721
Number analyzed (Participants) | 10 | 10 | 9
nanograms/milliliter (ng/mL) | 183 (41) | 180 (17) | 888 (11)

3. Primary Outcome: Pharmacokinetics: Area Under the Curve Extrapolated to Infinity (AUC0-∞) of Cerebrospinal Fluid (CSF) LY2886721
Description: AUC0-∞ following administration of a single dose of 70 mg LY2886721.
Time Frame: Predose through 36 hours after administration of study drug
Population: Participants who received at least one dose of LY2886721 at the 70-mg dose level and with evaluable CSF LY2886721-concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort B: 70 mg LY2886721
Number analyzed (Participants) | 10 | 10
ng*h/mL | 458 (16) | 410 (16)

4. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of CSF LY2886721
Description: Cmax following administration of a single dose of 70 mg LY2886721.
Time Frame: Predose through 36 hours after administration of study drug
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Cohort A: 70 mg LY2886721: Participants with Alzheimer's received a single, 70-mg (1 capsule), oral dose of LY2886721.
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort B: 70 mg LY2886721
Number analyzed (Participants) | 10 | 10
ng/mL | 24.0 (18) | 24.4 (19)

5. Primary Outcome: Pharmacodynamics (PD): Cnadir of Plasma Amyloid β (Aβ)1-40
Description: Plasma concentration of Aβ1-40 was summarized based on lowest observed concentration (Cnadir).
Time Frame: Predose, up to 96 hours after administration of study drug
Population: Participants who received at least one dose of LY2886721 or placebo and had evaluable plasma Aβ 1-40 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms/milliliter (pg/mL)
Groups:
- Cohorts B and C: Placebo: Healthy participants received a single, oral dose of LY2886721-matching placebo (1 capsule).
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort A: Placebo | Cohort B: 70 mg LY2886721 | Cohort C: 280 mg LY2886721 | Cohorts B and C: Placebo
Number analyzed (Participants) | 10 | 2 | 10 | 9 | 5
picograms/milliliter (pg/mL) | 22.2 (35.2) | 140 (NA) — Geometric Coefficient of Variation not reported since n <3. | 19.5 (11.9) | 11.0 (42.2) | 162 (7.39)

6. Primary Outcome: PD: Cnadir of CSF Aβ 1-40
Description: Plasma concentration of Aβ1-40 was summarized based on Cnadir following administration of a single dose of 70 mg LY2886721 or a single dose of LY2886721-matching placebo.
Time Frame: Predose up to 36 hours after administration of study drug
Population: Participants who received at least one dose of LY2886721 at the 70-mg dose level or placebo and had evaluable CSF Aβ 1-40 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- Cohort A: Placebo: Participants with Alzheimer's received a single, oral dose of LY2886721-matching placebo (1 capsule).
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort A: Placebo | Cohort B: 70 mg LY2886721 | Cohort B: Placebo
Number analyzed (Participants) | 10 | 2 | 10 | 2
pg/mL | 7600 (30.7) | 19500 (NA) — Geometric Coefficient of Variation not reported since n <3. | 4480 (110) | 12500 (NA) — Geometric Coefficient of Variation not reported since n <3.

7. Secondary Outcome: Cohort C: Mean QTcF Value at Cmax
Description: The mean QTcF value at Cmax for participants administered a single dose of 280 mg LY2886721 was reported. The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. Time matched mean change from baseline in QTcF = time matched plasma concentration + participant + random error.
Time Frame: Predose up to 48 hours after administration of study drug
Population: Participants who received at least one dose of LY2886721 at the 280-mg dose level and with evaluable mean QTcF data.
Measure: Mean (90% Confidence Interval); unit: milliseconds (ms)
Arm/Group | Cohort C: 280 mg LY2886721
Number analyzed (Participants) | 9
milliseconds (ms) | 28.3 [23.4 to 33.2]

ADVERSE EVENTS:
Arm/Group | Cohort A: 70 mg LY2886721 | Cohort A: Placebo | Cohort B: 70 mg LY2886721 | Cohort B: Placebo | Cohort C: 280 mg LY2886721 | Cohort C: Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/2 | 0/10 | 0/2 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 4/10 | 1/2 | 8/10 | 0/2 | 1/9 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: 70 mg LY2886721 (N=10) | Cohort A: Placebo (N=2) | Cohort B: 70 mg LY2886721 (N=10) | Cohort B: Placebo (N=2) | Cohort C: 280 mg LY2886721 (N=9) | Cohort C: Placebo (N=3)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Red blood cells csf positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (2) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days